CLINICAL TRIAL: NCT03346694
Title: Reducing Surgical Site Infection Rates Using an Alternative Sternal Dressing
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jack Boyd, Prinicipal Investigator, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 41985
Record Dates: First submitted 2017-11-15; First posted 2017-11-17 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Wound of Skin

STUDY DESIGN:
Intervention Model Description: Participant randomly assigned to either a control or one of two intervention groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Dressing 1: Standard Island Dressing (Active Comparator): Standard dressing that is applied on most patients with a sternotomy wound incision immediately after cardiovascular surgery before leaving the operating room. Dressing will be removed 48 hours after surgery.
  Interventions: Device: Standard Island Dressing
- Dressing 2: Prevena negative pressure (Active Comparator): Prevena negative pressure wound suction machine dressing applied to sternotomy wound incision immediately after cardiovascular surgery. Dressing will be in use for 7 days or removed sooner if participant is discharged before end of 7 day post-operative time period.
  Interventions: Device: Prevena Negative Pressure wound dressing
- Dressing 3: Mepilex Border Post-Op Ag (Active Comparator): Mepilex Border PostOp AG dressing impregnated with silver ions. Dressing will be in use for 7 days or removed earlier if patient is discharged before end of 7 days post0operative time period.
  Interventions: Device: Mepilex Border Post-Op Ag

INTERVENTIONS:
Device: Standard Island Dressing — participant randomized to control group before end of surgery to be applied on cardiovascular heart surgical sternal incision.
  Other Names: Dressing 1
  Arms: Dressing 1: Standard Island Dressing
Device: Prevena Negative Pressure wound dressing — participant randomized to dressing before end of surgery to be applied on cardiovascular heart surgical sternal incision.
  Other Names: Dressing 2
  Arms: Dressing 2: Prevena negative pressure
Device: Mepilex Border Post-Op Ag — Participant randomized to dressing before end of surgery to be applied on cardiovascular heart surgical sternal incision
  Other Names: Dressing 3
  Arms: Dressing 3: Mepilex Border Post-Op Ag

SUMMARY:
This study will evaluate two alternative dressings compared to a standard Island dressing presently in use at Stanford Hospital to determine reductions in surgical site infection (SSI) rates among cardiac surgery patients. Cardiovascular surgery patients who will have a sternotomy incision as a routine part of their surgery will be approached to voluntarily participate. Participants will be randomized to one of three dressing to determine which dressing has the lowest rate of sternal wound infection. The investigators will also assess the impact of alternative dressing use on hospital 30-day readmission rates related to SSI.

ELIGIBILITY:
Inclusion Criteria:

* Participants who will undergo cardiac surgery via a sternotomy incision.Inclusion criteria will be patients having surgical valve, CABGs, aortic dissection, myectomy and myotomy, Cox MAZE, Myocardial bridge Un-roofing

Exclusion Criteria:

* Patients undergoing heart transplants, Ventricular Assist Device (VAD), with postoperative courses complicated by tamponade, take-backs, and open chest incisions will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 660 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2030-05-01 (Estimated); Study Completion 2035-05-01 (Estimated)

PRIMARY OUTCOMES:
Rates of surgical site infection pertaining to each dressing studied. | From Post-Operative date 0 to 7th day or earlier which ever day comes first.
  evaluate alternative dressings to determine reductions in surgical site infection (SSI) rates among cardiac surgery patients

SECONDARY OUTCOMES:
Impact of alternative dressings on rates of Sternal wound incision infection | 30 days after participant discharge.
  Assess the impact of alternative dressing use on hospital 30-day readmission rates related to surgical site infection (SSI).

CONTACTS AND LOCATIONS:
Overall Officials: Jack Boyd, M.D., Principal Investigator — Cardiovascular Surgeon
Locations (1):
- Stanford Healthcare, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lwanga, S.K. & Lemeshow, S. (1991). Sample size determination in health studies: a practical manual. World Health Organization: Geneva, Switzerland.
- [Background] R Core Team (2016). R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria.
- [Result] Barnes S. What's new in SSI prevention? AORN J. 2015 Jun;101(6):P10-2. doi: 10.1016/s0001-2092(15)00421-4. No abstract available. PMID 26219113
- [Result] Ly, E. (2015). Cardiothoracic (CT) surgery data summary- all surgical site infections by quarter 2015 [PowerPoint slides]. Retrieved from personal communication.
- [Result] Kles CL, Murrah CP, Smith K, Baugus-Wellmeier E, Hurry T, Morris CD. Achieving and Sustaining Zero: Preventing Surgical Site Infections After Isolated Coronary Artery Bypass With Saphenous Vein Harvest Site Through Implementation of a Staff-Driven Quality Improvement Process. Dimens Crit Care Nurs. 2015 Sep-Oct;34(5):265-72. doi: 10.1097/DCC.0000000000000131. PMID 26244240
- See also: A Language and environment for statistical computing — https://www.R-project.org/